CLINICAL TRIAL: NCT05177367
Title: Combined Effects of Variety and Portion Size on Meal Intake of Women
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study design has changed.
Sponsor: Penn State University (Other)
Collaborators: Jenny Craig, Inc. (Industry)
Responsible Party: Principal Investigator, Barbara J. Rolls, Professor of Nutrition and Director of The Laboratory For The Study of Human Ingestive Behavior, Penn State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: FoodVariety102
Record Dates: First submitted 2021-12-15; First posted 2022-01-04 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Eating Behavior
MeSH Terms: conditions — Feeding Behavior | interventions — Food

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Sequential Variety, Small Portion (Experimental): 3 courses each consisting of a different food served in a small portion.
  Interventions: Other: Sequential Variety; Other: Small portion
- Sequential Variety, Large Portion (Experimental): 3 courses each consisting of a different food served in a large portion.
  Interventions: Other: Sequential Variety; Other: Large Portion
- Simultaneous Variety, Small Portion (Experimental): 3 courses each consisting of 3 foods served in small portions.
  Interventions: Other: Simultaneous Variety; Other: Small portion
- Simultaneous Variety, Large Portion (Experimental): 3 courses each consisting of 3 foods served in large portions.
  Interventions: Other: Simultaneous Variety; Other: Large Portion
- Single Food, Small Portion (Experimental): 3 courses each consisting of the same food served in a small portion.
  Interventions: Other: Single Food; Other: Small portion
- Single Food, Large Portion (Experimental): 3 courses each consisting of the same food served in a large portion.
  Interventions: Other: Single Food; Other: Large Portion

INTERVENTIONS:
Other: Sequential Variety — 3 courses each consisting of a different food
  Arms: Sequential Variety, Large Portion; Sequential Variety, Small Portion
Other: Simultaneous Variety — 3 courses each consisting of 3 foods
  Arms: Simultaneous Variety, Large Portion; Simultaneous Variety, Small Portion
Other: Single Food — 3 courses each consisting of the same food
  Arms: Single Food, Large Portion; Single Food, Small Portion
Other: Small portion — Small meal portion size
  Arms: Sequential Variety, Small Portion; Simultaneous Variety, Small Portion; Single Food, Small Portion
Other: Large Portion — Large meal portion size
  Arms: Sequential Variety, Large Portion; Simultaneous Variety, Large Portion; Single Food, Large Portion

SUMMARY:
The primary purpose of this study is to investigate the combined effects of meal variety and portion size on food intake at a meal. The study will also investigate relationships with eating microstructure such as eating rate and bite size. Additionally, other individual characteristics will be examined for their influence on the effects of variety and portion size on meal intake.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to travel to Penn State University Park campus weekly for meals
* Be fully vaccinated against COVID-19
* Be a woman 20 - 65 years old
* Regularly eat 3 meals/day
* Be willing to refrain from drinking alcohol the day before and during test days
* Have a body mass index between 18.0 and 35.0 kg/m*m
* Be willing to refrain from eating after 10 pm the evening before test sessions
* Be willing to participate in all study procedures

Exclusion Criteria:

* Must not be a smoker
* Must not be an athlete in training
* Must not be pregnant or breastfeeding at the time of screening
* Must not have taken prescription or non-prescription drugs that may affect appetite or food intake within the last 3 months
* Must not dislike or be unable to eat the test foods (because of allergies, intolerance, or dietary restrictions)
* Must not have a high variability in liking of the test foods
* Must not be currently dieting to gain or lose weight
* Must not have a health condition that affects appetite
* Must not have participated in a similar study in our lab in the past year
* Must not be a student, faculty, or staff member in nutritional sciences or psychology

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-02-20 (Estimated); Primary Completion 2023-01-20 (Estimated); Study Completion 2023-01-27 (Estimated)

PRIMARY OUTCOMES:
Change in intake by weight | Weeks 1, 2, 3, 4, 5, 6
  Weight (grams) of all meal components consumed
Change in energy intake | Weeks 1, 2, 3, 4, 5, 6
  Energy intake (kilocalories) of all meal components consumed, calculated from weight and energy density

SECONDARY OUTCOMES:
Change in bite count | Weeks 1, 2, 3, 4, 5, 6
  The number of bites of food during the meal
Change in meal duration | Weeks 1, 2, 3, 4, 5, 6
  Duration of the meal in minutes
Change in mean eating rate | Weeks 1, 2, 3, 4, 5, 6
  Mean food intake per minute (grams/minute), calculated by dividing meal food intake by meal duration
Change in mean bite size | Weeks 1, 2, 3, 4, 5, 6
  Mean food intake per bite (grams/bite), calculated by dividing meal food intake by bite count
Change in sip count | Weeks 1, 2, 3, 4, 5, 6
  The number of sips of water during the meal
Change in mean drinking rate | Weeks 1, 2, 3, 4, 5, 6
  Mean water intake per minute (grams/minute), calculated by dividing meal water intake by meal duration
Change in mean sip size | Weeks 1, 2, 3, 4, 5, 6
  Mean water intake per sip (grams/sip), calculated by dividing meal water intake by sip count
Change in switching between bites and sips | Weeks 1, 2, 3, 4, 5, 6
  The number of switches between bites and sips during the meal
Change in switching between different foods | Weeks 1, 2, 3, 4, 5, 6
  The number of switches between different foods
Change in rating of pleasantness of the taste of food samples | From before the test meal to after the test meal in weeks 1, 2, 3, 4, 5, 6
  Measured on a 100-mm visual analogue scale ranging from not at all pleasant (0 mm) to extremely pleasant (100 mm). This will be used to calculate Sensory-Specific Satiety
Change in rating of prospective consumption of food samples | Time Frame: From before the test meal to after the test meal in weeks 1, 2, 3, 4, 5, 6
  Measured on a 100-mm visual analogue scale ranging from none at all (0 mm) to a very large amount (100 mm), in answer to "How much of [this food] do you want to eat right now?". This will be used to calculate Sensory-Specific Satiety
Change in rating of hunger | Time Frame: From before the test meal to after the test meal in weeks 1, 2, 3, 4, 5, 6
  Measured on a 100-mm visual analogue scale ranging from not at all hungry (0 mm) to extremely hungry (100 mm)
Change in rating of thirst | Time Frame: From before the test meal to after the test meal in weeks 1, 2, 3, 4, 5, 6
  Measured on a 100-mm visual analogue scale ranging from not at all thirsty (0 mm) to extremely thirsty (100 mm)
Change in rating of nausea | Time Frame: From before the test meal to after the test meal in weeks 1, 2, 3, 4, 5, 6
  Measured on a 100-mm visual analogue scale ranging from not at all nauseated (0 mm) to extremely nauseated (100 mm)
Change in rating of fullness | Time Frame: From before the test meal to after the test meal in weeks 1, 2, 3, 4, 5, 6
  Measured on a 100-mm visual analogue scale ranging from not at all full (0 mm) to extremely full (100 mm)

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratory for the Study of Human Ingestive Behavior, The Pennsylvania State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No